CLINICAL TRIAL: NCT01174329
Title: Difference in Salivary Flow in Patients With Salivary Gland Hypofunction of the Following Application of Neuro-electrostimulation
Brief Title: Treatment of Salivary Gland Hypofunction With Neuro- Electrostimulation
Acronym: SALELECTROSTIM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Dr Mario Cesar Salinas Carmona, Universidad Autónoma de Nuevo León
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2010-07-28; First posted 2010-08-03 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-07

CONDITIONS: Xerostomia; Polypharmacy; Sjögren's Syndrome
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient-regulated neuro-electrostimulation by "Saliwell Crown" (Experimental): Patient regulated (by a remote control) neuro-electrostimulation by "Saliwell Crown"
  Interventions: Device: Patient-regulated neuro-electrostimulation by "Saliwell Crown"
- Automatic neuro-electrostimulation by "Saliwell Crown" (Active Comparator): No remote control used
  Interventions: Device: Automatic neuro-electrostimulation by "Saliwell Crown"

INTERVENTIONS:
Device: Automatic neuro-electrostimulation by "Saliwell Crown" — Continuous stimulation of the lingual nerve by "Saliwell Crown"
  Arms: Automatic neuro-electrostimulation by "Saliwell Crown"
Device: Patient-regulated neuro-electrostimulation by "Saliwell Crown" — On-demand stimulation of the lingual nerveby "Saliwell Crown"
  Arms: Patient-regulated neuro-electrostimulation by "Saliwell Crown"

SUMMARY:
The objective of the study is to evaluate with clinical parameters the performance of Saliwell Crown as a neuro-electrostimulator of the submandibular and sublingual salivary glands in hypofunction status due to polypharmacy or Sjögren's Syndrome in patients with symptoms of xerostomia.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 75 years of age
* Clinical symptoms of xerostomia
* Difference in whole salivary flow between resting and stimulating conditions
* Patient ASA type I to III
* Absence of at least one mandibular third molar inferior, but at least partially dentated in the mandible

Exclusion Criteria:

* Patients with antimicrobial treatments in the three previous months
* Smokers
* Intake of bisphosphonates
* Limitation of mandibular opening
* Interoclusal distance smaller than 10 millimetres
* Lack of adequate bone availability for implant placement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
self-reported xerostomia | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- C.D. Especialidad de Periodoncia, Monterrey, Nuevo León, Mexico